CLINICAL TRIAL: NCT00325351
Title: Phase 1/2 Study of ZK-Epothilone (ZK-Epo; ZK-219477) in Combination With Carboplatin in Patients With Platinum-sensitive Recurrent Ovarian Cancer
Brief Title: ZK-Epo Given With Carboplatin in Patients With Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91476; 307979 (Other: company internal)
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Ovarian Neoplasms
Keywords: Ovarian cancer; Ovarian neoplasms, epithelium
MeSH Terms: conditions — Ovarian Neoplasms | interventions — sagopilone; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Sagopilone (ZK 219477) + carboplatin

INTERVENTIONS:
Drug: Sagopilone (ZK 219477) + carboplatin — Chemotherapy for recurrent ovarian cancer

SUMMARY:
The purpose of this study is to evaluate whether treatment with a new drug called ZK-Epothilone (ZK-Epo) given with carboplatin in patients with recurrent ovarian cancer, who previously have had a good response with cisplatin or carboplatin, is safe and helps to decrease or stop tumor growth.

DETAILED DESCRIPTION:
This study has previously been registered by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.Bayer HealthCare Pharmaceuticals, Inc. is sponsoring this trial.

ELIGIBILITY:
Inclusion Criteria:- Must have evidence of ovarian cancer measurable by computed tomography (CT) scan or by CA125 blood levels- No radiation therapy in last 4 weeks- No chemotherapy in last 24 weeks - No immunotherapy in last 4 weeks- Good response after previous treatment with carboplatin or cisplatin and then the ovarian cancer got worse again after at least 6 months- Additional criteria determined at screening visit Exclusion Criteria:- Having had more than one treatment regimen with carboplatin or cisplatin- Prior treatment with other epothilones (e.g. ixabepilone)- Use of any investigational drug in the last 4 weeks- Previous radiation to the whole pelvis- Symptomatic brain tumors requiring radiation to the brain - Active infection- Pregnant or breast feeding- Additional criteria determined at screening visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-08-24 (Actual); Primary Completion 2008-07-08 (Actual); Study Completion 2009-03-25 (Actual)

PRIMARY OUTCOMES:
Response to treatment with ZK-Epo after 6 cycles | After 6 cycles

SECONDARY OUTCOMES:
Safety and tolerability of ZK-Epo given with carboplatin | Sept. 2008

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (16):
- United States (14):
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Bakersfield, California
  - La Jolla, California
  - San Diego, California
  - Savannah, Georgia
  - South Bend, Indiana
  - Baltimore, Maryland
  - Albuquerque, New Mexico
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Knoxville, Tennessee
  - Roanoke, Virginia
- Canada (2):
  - Calgary, Alberta
  - Toronto, Ontario

REFERENCES:
- [Result] McMeekin S, Patel R, Verschraegen C, Celano P, Burke J 2nd, Plaxe S, Ghatage P, Giurescu M, Stredder C, Wang Y, Schmelter T. Phase I/II study of sagopilone (ZK-EPO) plus carboplatin in women with recurrent platinum-sensitive ovarian cancer. Br J Cancer. 2012 Jan 3;106(1):70-6. doi: 10.1038/bjc.2011.499. Epub 2011 Nov 22. PMID 22108514